CLINICAL TRIAL: NCT03355716
Title: Post-operative Pain Relief in Laparoscopic Cholecystectomy Using a Combination of Intraperitoneal Bupivacaine Morphine, Bupivacaine Fentanyl and Bupivacaine Ketamine: A Comparative Study
Brief Title: Post-operative Pain Relief in Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Mahmoud, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: post-oprative pain relief
Record Dates: First submitted 2017-11-21; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Morphine; Fentanyl; Ketamine

STUDY DESIGN:
Intervention Model Description: At the end of the procedure, all the subjects will be randomly allocated to groups using computer-generated random numbers. Each group of 30 subjects, that is,
  Group A (placebo):
  instillation of bupivacaine alone: Bupivacaine 25 ml (0.25%) after surgery completion;
  Group B :
  Instillation of bupivacaine and morphine: Bupivacaine 25 ml (0.25%) + Morphine (3.0 mg)
  Group C :
  Instillation of bupivacaine and fentanyl: Bupivacaine25 ml (0.25%) + fentanyl (30.0 Mc)
  Group D :
  Instillation of bupivacaine and Ketamine: Bupivacaine25 ml (0.25%) + ketamine (0.5 mg/kg).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (placebo): (Placebo Comparator): instillation of bupivacaine alone: Bupivacaine 25 ml (0.25%) after surgery completion
  Interventions: Drug: bupivacaine
- Group B (Active Comparator): Instillation of bupivacaine and morphine: Bupivacaine 25 ml (0.25%) + Morphine (3.0 mg)
  Interventions: Drug: bupivacaine; Drug: morphine
- Group C (Active Comparator): Instillation of bupivacaine and fentanyl: Bupivacaine25 ml (0.25%) + fentanyl (30.0 Mc)
  Interventions: Drug: bupivacaine; Drug: fentanyl
- Group D (Active Comparator): Instillation of bupivacaine and Ketamine: Bupivacaine25 ml (0.25%) + ketamine (0.5 mg/kg).
  Interventions: Drug: bupivacaine; Drug: Ketamine:

INTERVENTIONS:
Drug: bupivacaine — Bupivacaine 25 ml (0.25%)
Drug: morphine — Morphine (3.0 mg)
  Arms: Group B
Drug: fentanyl — fentanyl (30.0 Mc)
  Arms: Group C
Drug: Ketamine: — ketamine (0.5 mg/kg).
  Arms: Group D

SUMMARY:
compare the analgesic efficacy of the combination of bupivacaine and morphine, bupivacaine and fentanyl and bupivacaine and ketamine in alleviating post operative pain following laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is comparatively advantageous over open cholecystectomy in pain management with shorter duration of hospital stays. Pain management is medically pertinent for optimal care in surgical patients. Although development and advancement in understanding of the patho-physiology of pain, analgesics, pharmacology and the development of better effective techniques for post-operative pain control, patients still continue to experience considerable discomfort.

Laparotomy results in parietal pain, whereas laparoscopy has a visceral component, a somatic component and shoulder pain secondary to diaphragmatic irritation because of CO2 pneumo-peritoneum. Postoperative pain associated with laparoscopic cholecystectomy, although less severe and of shorter duration than that after open cholecystectomy, is still a source of marked discomfort and surgical stress. The degree of the pain after laparoscopic procedures has multifactorial influence including the volume of residual gas, type of gas used for pneumo-peritoneum, pressure created by the pneumo-peritoneum and insufflated gas temperature.

Local anesthetic infiltration of the incision sites decreases postoperative opiate requirement and improves subjective pain scores but does eliminate the pain.

Earlier scientists have also reported several beneficial effects of the intra-peritoneal application of bupivacaine with morphine on postoperative pain management after laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I and II
* scheduled for elective laparoscopic cholecystectomy
* under a standardized general anesthesia technique.

Exclusion Criteria:

* uncooperative, unwilling,
* history of anaphylaxis to local anesthetics and/or opioids and the drugs to be used,
* history of drug abuse,
* anmorbidly obese patients,
* ASA classification III, IV, V
* d patients having any other significant co-morbidities
* any other with psychiatric disease
* pregnant women

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
post operative pain | 24 hours
  All subjects will be familiar with the visual analogue scale of pain (VAS) score preoperatively and will be instructed in detail on its use as a tool for measuring postoperative pain The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme .
  A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in postsurgical patients (knee replacement, hysterectomy, or laparoscopic myomectomy) who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm) .

REFERENCES:
- [Background] Khurana S, Garg K, Grewal A, Kaul TK, Bose A. A comparative study on postoperative pain relief in laparoscopic cholecystectomy: Intraperitoneal bupivacaine versus combination of bupivacaine and buprenorphine. Anesth Essays Res. 2016 Jan-Apr;10(1):23-8. doi: 10.4103/0259-1162.164731. PMID 26957685